CLINICAL TRIAL: NCT00409448
Title: Improving Mental Health Outcomes of Child Brain Injury
Brief Title: Internet-Based Treatment for Children With Traumatic Brain Injuries & Their Families: Counselor Assisted Problem Solving
Acronym: CAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH073764 (NIH); DDTR B2-NDA
Record Dates: First submitted 2006-12-07; First posted 2006-12-08 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Traumatic Brain Injury
Keywords: TBI; intracranial edema; brain edema; craniocerebral trauma; head injury; brain hemorrhage, traumatic; subdural hematoma; brain concussion; head injuries, closed; epidural hematoma; extra-axial hemorrhage; cortical contusion
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Edema; Craniocerebral Trauma; Brain Hemorrhage, Traumatic; Hematoma, Subdural; Brain Concussion; Head Injuries, Closed; Hematoma, Epidural, Spinal; Brain Contusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CAPS (Experimental): Participants will receive the Internet-based counselor-assisted problem-solving group treatment
  Interventions: Behavioral: Counselor-assisted problem solving (CAPS)
- IRC (Active Comparator): Participants will receive the Internet resource comparison group treatment
  Interventions: Behavioral: Internet-resource comparison (IRC)

INTERVENTIONS:
Behavioral: Counselor-assisted problem solving (CAPS) — In CAPS, a trained counselor will guide families through a 6-month structured online problem-solving and skill-building program via one-on-one videoconference sessions.
  Arms: CAPS
Behavioral: Internet-resource comparison (IRC) — Families in the IRC group will receive computers, high speed internet access, and links to brain injury information and resources, but not the CAPS website content.
  Arms: IRC

SUMMARY:
This study will evaluate the effectiveness of an Internet-based psychosocial treatment in improving problem-solving, communication skills, stress management strategies, and coping among children who have had a traumatic brain injury and their families.

DETAILED DESCRIPTION:
A traumatic brain injury (TBI) is caused by a strong blow, jolt, or penetration to the head that disrupts normal brain functioning. A TBI can range from a mild concussion to severe brain damage. Falls, assaults, and motor vehicle accidents account for more than 50% of TBIs. Physical symptoms of a TBI can be subtle to severe and can include nausea, memory loss, mood swings, blurred vision, and light-headedness. This type of injury can be very stressful for families and can result in feelings of anxiety, burden, and depression among family members. A child who experiences a TBI will often display new social and behavioral problems, leading to further parental distress and increased family dysfunction. Recent studies have shown that problem-solving interventions can reduce caregiver distress and improve child adjustment following a TBI. However, access to skilled therapists and specialized care for this kind of psychosocial treatment is often limited in many communities. In such communities, the Internet offers a new way to meet the mental and other health needs of individuals with TBIs. This study will evaluate the effectiveness of an Internet-based psychosocial treatment in improving problem solving, communication skills, stress management strategies, and coping among teens who have had a TBI and their families.

Families participating in this study will be randomly assigned to either an Internet-based counselor-assisted problem-solving (CAPS) group or an Internet resource comparison group (IRC). Participants assigned to CAPS will work with a trained counselor who will guide them through a 6-month structured online problem-solving and skill-building program via one-on-one videoconference sessions. Families assigned to IRC will receive computers, high speed Internet access, and links to brain injury information and resources, but no access to the CAPS Web site content. The effectiveness of CAPS will be assessed after treatment and at 6- and 12-month follow-up evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe TBI that occurred within the last 6 months
* Overnight hospital stay
* English-speaking
* Parent must be willing to provide informed consent

Exclusion Criteria:

* Child does not live with parents or guardian
* Child or parent has history of hospitalization for psychiatric problem
* TBI is a result of child abuse
* Child suffered a nonblunt injury (e.g., projectile wound, stroke, drowning, or other form of asphyxiation)
* Diagnosed with moderate or severe mental retardation, autism, or a significant developmental disability

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 132 (Actual)
Dates: Start 2007-03; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Parent report measures | 5 years
Teen self-report measures | 5 years

SECONDARY OUTCOMES:
Neuropsychological testing | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Shari L. Wade, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (5):
- United States (5):
  - Denver Children's Hospital, Denver, Colorado
  - The Mayo Clinic, Rochester, Minnesota
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio

REFERENCES:
- [Derived] Narad ME, Kaizar EE, Zhang N, Taylor HG, Yeates KO, Kurowski BG, Wade SL. The Impact of Preinjury and Secondary Attention-Deficit/Hyperactivity Disorder on Outcomes After Pediatric Traumatic Brain Injury. J Dev Behav Pediatr. 2022 Aug 1;43(6):e361-e369. doi: 10.1097/DBP.0000000000001067. Epub 2022 Feb 15. PMID 35170571
- [Derived] Wade SL, Kaizar EE, Narad M, Zang H, Kurowski BG, Yeates KO, Taylor HG, Zhang N. Online Family Problem-solving Treatment for Pediatric Traumatic Brain Injury. Pediatrics. 2018 Dec;142(6):e20180422. doi: 10.1542/peds.2018-0422. Epub 2018 Nov 9. PMID 30413559
- [Derived] Huebner ARS, Cassedy A, Brown TM, Taylor HG, Stancin T, Kirkwood MW, Wade SL. Use of Mental Health Services by Adolescents After Traumatic Brain Injury: A Secondary Analysis of a Randomized Controlled Trial. PM R. 2018 May;10(5):462-471. doi: 10.1016/j.pmrj.2017.10.004. Epub 2017 Oct 31. PMID 29097272
- [Derived] Narad ME, Minich N, Taylor HG, Kirkwood MW, Brown TM, Stancin T, Wade SL. Effects of a Web-Based Intervention on Family Functioning Following Pediatric Traumatic Brain Injury. J Dev Behav Pediatr. 2015 Nov-Dec;36(9):700-7. doi: 10.1097/DBP.0000000000000208. PMID 26461100
- [Derived] Wade SL, Taylor HG, Cassedy A, Zhang N, Kirkwood MW, Brown TM, Stancin T. Long-Term Behavioral Outcomes after a Randomized, Clinical Trial of Counselor-Assisted Problem Solving for Adolescents with Complicated Mild-to-Severe Traumatic Brain Injury. J Neurotrauma. 2015 Jul 1;32(13):967-75. doi: 10.1089/neu.2014.3684. Epub 2015 May 7. PMID 25738891
- [Derived] Wade SL, Kurowski BG, Kirkwood MW, Zhang N, Cassedy A, Brown TM, Nielsen B, Stancin T, Taylor HG. Online problem-solving therapy after traumatic brain injury: a randomized controlled trial. Pediatrics. 2015 Feb;135(2):e487-95. doi: 10.1542/peds.2014-1386. Epub 2015 Jan 12. PMID 25583911
- [Derived] Kurowski BG, Wade SL, Kirkwood MW, Brown TM, Stancin T, Taylor HG. Long-term benefits of an early online problem-solving intervention for executive dysfunction after traumatic brain injury in children: a randomized clinical trial. JAMA Pediatr. 2014 Jun;168(6):523-31. doi: 10.1001/jamapediatrics.2013.5070. PMID 24781374
- [Derived] Arnett AB, Peterson RL, Kirkwood MW, Taylor HG, Stancin T, Brown TM, Wade SL. Behavioral and cognitive predictors of educational outcomes in pediatric traumatic brain injury. J Int Neuropsychol Soc. 2013 Sep;19(8):881-9. doi: 10.1017/S1355617713000635. Epub 2013 Jun 21. PMID 23790158
- [Derived] Kurowski BG, Wade SL, Kirkwood MW, Brown TM, Stancin T, Taylor HG. Online problem-solving therapy for executive dysfunction after child traumatic brain injury. Pediatrics. 2013 Jul;132(1):e158-66. doi: 10.1542/peds.2012-4040. Epub 2013 Jun 10. PMID 23753094
- [Derived] Wade SL, Stancin T, Kirkwood M, Brown TM, McMullen KM, Taylor HG. Counselor-assisted problem solving (CAPS) improves behavioral outcomes in older adolescents with complicated mild to severe TBI. J Head Trauma Rehabil. 2014 May-Jun;29(3):198-207. doi: 10.1097/HTR.0b013e31828f9fe8. PMID 23640543